CLINICAL TRIAL: NCT01735942
Title: A Comparison of Ingenol Mebutate and Cryotherapy for Treatment of Actinic Keratoses.
Brief Title: Ingenol Mebutate Compared to Cryotherapy for the Treatment of Skin Lesions
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU68227
Record Dates: First submitted 2012-11-05; First posted 2012-11-28 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ingenol Mebutate (Experimental): Ingenol Mebutate applied to one side of face with skin lesions
  Interventions: Drug: Ingenol mebutate
- Cryotherapy (Active Comparator): Cryotherapy applied to other side of face with skin lesions
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Drug: Ingenol mebutate
  Arms: Ingenol Mebutate
Procedure: cryotherapy
  Arms: Cryotherapy

SUMMARY:
The purpose of this study is to find out the effectiveness of ingenol mebutate compared to cryotherapy (freezing of the tissue) for the treatment of face and scalp skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 89 years old.
* Have at least a total of 10 non-hypertrophic actinic keratoses (AKs) on the face and scalp
* The subjects are in good health
* The subjects have the willingness and the ability to understand and provide informed consent for the use of their tissue and are able to communicate with the investigator

Exclusion Criteria:

* Subjects under 18 years of age and over the age of 89
* Subjects who are pregnant or lactating
* Subjects with sensitivity to cold
* Subjects with use of topical medications such as corticosteroids, alpha-hydroxyacids or retinoids 2 weeks before study entry
* Subjects who received previous treatment of target AKs
* Subjects whose target treatment area was within 5 cm of an incompletely healed wound or within 10 cm of a suspected basal-cell or squamous-cell carcinoma
* Subjects with use of medications or other treatments that could interfere with evaluation of the treatment area within 2 months before study entry (e.g., topical medications, artificial tanners, immunosuppressive medications, immunomodulating agents, cytotoxic drugs, ultraviolet B phototherapy, other therapies for actinic keratoses, or oral retinoids)
* Subjects who are unable to understand the protocol or to give informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual assessment scores at 3 months | Baseline and 3 months
  The visual assessment evaluates seven clinical signs: erythema, edema, wheal vesiculation, ulceration, hemorrhage, purpura, and crusting. Each sign is assigned a score of 0 to 3, where a score of 0 is associated with no expression of the clinical sign and a better outcome, and a score of 3 is associated with severe expression of the clinical sign and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University